CLINICAL TRIAL: NCT05687500
Title: Oral Glibenclamide in Preterm Infants With Hyperglycaemia (GALOP)
Acronym: GALOP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160916J; 2021-005766-18 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2023-01-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Transient; Hypoglycemia, Neonatal; Preterm; Glibenclamide Adverse Reaction
Keywords: transient hypoglycemia; preterm; glibenclamide
MeSH Terms: conditions — Hypoglycemia; Premature Birth | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glibenclamide oral (Experimental): Amglidia®: glibenclamide oral suspension 6 mg/ml administered by gastric tube after dilution to 1/6th in human milk
  Interventions: Drug: Glibenclamide; Biological: Pharmacokinetics study; Biological: C-peptide proinsulin ratio; Biological: Routine biological monitoring

INTERVENTIONS:
Drug: Glibenclamide — Amglidia®: glibenclamide oral suspension 6 mg/ml administered by gastric tube after dilution to 1/6th in human milk
Biological: Pharmacokinetics study — * For the first 10 patients during the test phase, four 0.2 ml samples will be taken at H3, H6, H10, and H24 (+/- 1 hour) after the first dose; an additional sample will be taken for patients whose blood sugar levels stabilize beyond 24 hours, after 6 hours of stable blood sugar levels (4-10 mmol/l);
  * For subsequent patients included during phase II:
  * 1 sample of 0.2 ml within the first 24 hours of treatment, during a care assessment.
  * 1 sample of 0.2 ml within the first 24 hours of treatment, during a care assessment
  * 1 sample of 0.2 ml per day at each daily check-up as part of care during the treatment period.
  * In centers that are unable to perform the samples and the appropriate techniques for centralizing these PK points, these samples will not be taken.
  PK parameters of glibenclamide will be determined using nonlinear analysis: area under the plasma concentration time curve (AUC), absorption constant, apparent clearance and volume of distribution.
Biological: C-peptide proinsulin ratio — blood sampling at before first administration and after 24 hours for measurement of C-peptide proinsulin ratio if it is impossible to collect both volumes, the C-peptide collection will be prioritized
Biological: Routine biological monitoring — If there are not performed as part of standard care, biological monitoring of ALT, AST, complete blood count, hemostasis, urea, creatinine, blood ionogram, total bilirubin and conjugated bilirubin will be done before first administration at the following time frame : 48 hours after the first administration than each days during treatment period, and 48 hours after the end of treatment.
  Transaminases and hemostasis will be done only in case of clinical indication before the first administration.

SUMMARY:
The purpose of this study is to confirm hypothesis that Glibenclamide can be administered orally and is an alternative to insulin therapy in treating transient hyperglycemia of premature newborns.

DETAILED DESCRIPTION:
Transient hyperglycemia of premature newborns results from an overall decrease in insulin sensitivity, which is responsible at the beta cell level for abnormalities of intragranular cleavage of proinsulin into insulin, leading to reduced active insulin secretion. Intravenous administration of exogenous insulin can be used to combat insulin resistance and lower blood glucose, but it is difficult to manage in premature newborns and is associated with a substantial risk of hypoglycemia. Glibenclamide, which stimulates endogenous insulin secretion and can be administered orally, might be an alternative to insulin therapy in treating transient hyperglycemia of premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborn less than 34 week of amenorrhea corrected age
* Birth weight < 1500 g
* Birth term < 32 week of amenorrhea
* Hyperglycemia ≥ 10 mmol/l in 2 measurements, 3 hours apart after potential reduction of glucose intakes following each department's protocol
* Secure venous access point (umbilical venous catheter or epicutaneo-cava catheter)
* Enteral feeding considered before inclusion or already established
* Consent obtained from persons holding parental authority
* Beneficiary of social security

Exclusion Criteria

* Contraindication to enteral feeding (at the discretion of the clinician responsible for the child)
* Contraindication to glibenclamide according to current SPC
* Foetal growth restriction (FGR) birth weight < 3rd percentile (AUDIPOG definition)
* Severe birth defect, including cardiac malformation associated with a risk of myocardial ischemia
* Severe sepsis requiring mechanical ventilation or haemodynamic support
* Severe renal dysfunction (serum creatinine > 120 µmol/l)
* Severe hepatocellular failure (V factor less than the standard laboratory range for the age) and/or severe cholestasis (> 50 µmol/L)
* Hyperglycemia associated with an error in administering glucose infusion
* Profound hypophosphoremia (< 1 mmol/l)
* Hypersensitivity to glibenclamide or other sulphonylureas or sulphonamides, or one of the excipients
* Patient with continuous insulin IV administration
* Patient treated with miconazole

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Blood glucose control | At 72 hours after the first administration
  The primary evaluation criteria is 72 hours blood glucose control on glibenclamide treatment (success of the treatment). This is defined as the non-use of insulin and absence of severe hypoglycemia (< 1.5 mmol/l) or persistent moderate hypoglycemia (< 2.6 mmol/l in 2 successive measurements (dextro) at an interval of more than 3 hours)

SECONDARY OUTCOMES:
Overall success of the treatment | At 36 week of amenorrhea corrected age
  Overall success of the treatment defined by continuation to the end of treatment without recourse to insulin.
Blood glucose profile on glibenclamide | At the end of treatment assessed up to 15 days
  Time between the start of glibenclamide treatment and the 1st blood glucose < 10 mmol/l
Blood glucose profile on glibenclamide | At the end of treatment assessed up to 15 days
  Time between the start of glibenclamide treatment and the 1st blood glucose < 8 mmol/l
Blood glucose profile on glibenclamide | At the end of treatment assessed up to 15 days
  Proportion of time spent within the target blood glucose range (≥ 4 and < 10 mmol/l) during the period of glibenclamide treatment
Blood glucose profile on glibenclamide | At the end of treatment assessed up to 15 days
  Proportion of time spent above the target level (≥ 10 mmol/l) during the period of glibenclamide treatment
Blood glucose profile on glibenclamide | At the end of treatment assessed up to 15 days
  Proportion of time spent in hypoglycemia (< 2.6 mmol/l) during the period of glibenclamide treatment
Duration of glibenclamide treatment | At the end of treatment assessed up to 15 days
  Duration of glibenclamide treatment.
Nutritional intakes and growth | At the end of treatment assessed up to 15 days
  Carbohydrate
Nutritional intakes and growth: | At the end of treatment assessed up to 15 days
  lipid
Nutritional intakes and growth: | At the end of treatment assessed up to 15 days
  protein
Nutritional intakes and growth: | At the end of treatment assessed up to 15 days
  mean caloric intake (kcal/kg/day) during treatment
Nutritional intakes and growth: | At the end of treatment assessed up to 15 days
  mean weight gain (g/kg/day)
Nutritional intakes and growth | At 36 week of amenorrhea corrected age
  Carbohydrate
Nutritional intakes and growth: | At 36 week of amenorrhea corrected age
  lipid
Nutritional intakes and growth: | At 36 week of amenorrhea corrected age
  protein
Nutritional intakes and growth: | At 36 week of amenorrhea corrected age
  mean caloric intake (kcal/kg/day) during treatment
Nutritional intakes and growth: | At 36 week of amenorrhea corrected age
  mean weight gain ((g/kg/day)
Number of children with episode of hypoglycemia | At 72 hours after first administration
  Number of children with at least one episode of moderate (blood glucose < 2.6 mmol/l) or severe (< 1.5 mmol/l) hypoglycemia
Number of children with episode of hypoglycemia | At the end of treatment assessed up to 15 days
  Number of children with at least one episode of moderate (blood glucose < 2.6 mmol/l) or severe (< 1.5 mmol/l) hypoglycemia
Type of adverse reactions on glibenclamide | At 36 week of amenorrhea corrected age
  evaluation of the type of adverse reactions identified during the study
Number of adverse reactions on glibenclamide | At 36 week of amenorrhea corrected age
  evaluation of number of adverse reactions identified during the study
Number of participants with co-morbidity | At 36 week of amenorrhea corrected age
  Neonatal morbidity assessed at 36 WA corrected age: intraventricular haemorrhage, periventricular leukomalacia, retinopathy of premature newborns, haemodynamic disorders, ulcerative necrotising enterocolitis
Mortality | At 36 week of amenorrhea corrected age
  Mortality will be assessed
Dose adjustment | At the end of treatment assessed up to 15 days
  Number of dose adjustments, to evaluate the easy of use
ease of use by caregivers | At day one of treatment
  Assessment scores by visual-analogue scale for ease of use by caregivers; 0 as the lowest score, 10 as the highest score
ease of use by caregivers | At day two of treatment
  Assessment scores by visual-analogue scale for ease of use by caregivers; 0 as the lowest score, 10 as the highest score
ease of use by caregivers | At day three of treatment
  Assessment scores by visual-analogue scale for ease of use by caregivers; 0 as the lowest score, 10 as the highest score
Plasma concentrations of glibenclamide | At 3 hours after the first administration
  Evaluated by the pharmacokinetics study
Plasma concentrations of glibenclamide | At 6 hours after the first administration
  Evaluated by the pharmacokinetics study
Plasma concentrations of glibenclamide | At 10 hours after the first administration
  Evaluated by the pharmacokinetics study
Plasma concentrations of glibenclamide | At 24 hours after the first administration
  Evaluated by the pharmacokinetics study
Plasma concentrations of glibenclamide | At 24 hours of blood glucose stabilization
  Evaluated by the pharmacokinetics study

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BELTRAND, Pr, Study Director — Assistance Publique - Hôpitaux de Paris; Michel POLAK, Study Director — Assistance Publique - Hôpitaux de Paris; Delphine MITANCHEZ, Study Director — CHRU de Tours
Locations (1):
- Hopital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No